CLINICAL TRIAL: NCT01479205
Title: Security of the Bronchial Allergen Provocation With Mite and Aspergillus and Predictors for a Positive Reaction.
Brief Title: Induction of Allergen Specific Bronchial Immunotolerance After Specific Immunotherapy
Acronym: ITASIT
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Zielen, Prof. Dr. med Stefan Zieln, Johann Wolfgang Goethe University Hospital
Other Study IDs: FRAITASIT
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Mite Allergy; Allergic Asthma
Keywords: specific immunotherapy; bronchial allergen provocation; specific IgE; specific IgG; specific IgG4; SIT

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- mite allergic patients without SIT: patients suffering from allergic asthma/ rhino-conjunctivitis denying specific immunotherapy
- mite allergic patients with SIT: patients suffering from allergic asthma/ rhino-conjunctivitis undergoing mite specific immunotherapy

SUMMARY:
One aim of this study was to find out if the bronchial allergen provocation (BAP) is an appropriate method to appraise the efficacy of a specific immunotherapy (SIT). The investigators had one group of children receiving SIT and one group of patients who denied a SIT although they had an indication for it. Retrospectively the investigators analysed the data of the first BAP and blood parameters specific IgE-mite, total IgE before SIT (November 2008 till February 2010). Prospectively The investigators analysed the lung parameters and allergic labor parameters that we got in the course of the second BAP. The investigators mean parameter was PD20FEV1-mite. Another aim of The investigators study was to find specific immunological differences between children who improved because of SIT and those who showed no improvement. Thus, The investigators compared the levels of total IgE, cumulative IgE-mite and specific IgE-mite before and after SIT and the levels of specific IgG-mite and specific IgG4-mite after SIT.

DETAILED DESCRIPTION:
One aim of this study was to find out if the bronchial allergen provocation(BAP) is an appropriate method to appraise the efficacy of a specific immunotherapy (SIT). We had one group of children receiving SIT and one group of patients who denied a SIT although they had an indication for it. Retrospectively we analysed the data of the first BAP (PD20FEV1, VC, FEV1, FEV1/VC (%), eNO) and allergic blood parameters like specific IgE-mite, total IgE, cumulative IgE before SIT (November 2008 till February 2010). Prospectively we analysed the lung parameters and allergic labor parameters that we got in the course of the second BAP. Our mean parameter was PD20FEV1-mite. Another aim of our study was to find specific immunological differences between children who improved because of SIT and those who showed no improvement. Thus, we compared the levels of total IgE, cumulative IgE-mite and specific IgE-mite before and after SIT and the levels of specific IgG-mite and specific IgG4-mite after SIT. Additionally all patients answered a questionnaire according to ISAAC about their clinical symptoms, their quality of life and their medication score.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* between 5 and 18 years of age
* diagnosis of a moderate Asthma bronchiale (I-II) in the last 12 months or rhino conjunctivitis
* no exacerbation > 4 weeks before Visit

Exclusion Criteria:

* age < 5 years > 18 years,
* FEV1 < 75%
* no cooperation to undergo the BAP,
* exacerbation within the last 28 days before Visit
* other serious illnesses
* taking part in other clinical trials < 30 days

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 6-17 years of age with house dust mite allergy
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
improvement in BAP | one year after initiation of SIT
  significant improvement of PD20FEV1-mite in BAP

SECONDARY OUTCOMES:
Improvement of quality of life and medication | 1 year after initiation of SIT
  Via questionnaire (adapted from ISAAC-study) we assessed the quality of life, clinical symptoms and medication scores of the patients included

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof., Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Department of Paediatric Allergy and Pulmonology, Frankfurt am Main, Germany

REFERENCES:
- [Background] Abramson MJ, Puy RM, Weiner JM. Injection allergen immunotherapy for asthma. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD001186. doi: 10.1002/14651858.CD001186.pub2. PMID 20687065
- [Background] Pfaar O, Robinson DS, Sager A, Emuzyte R. Immunotherapy with depigmented-polymerized mixed tree pollen extract: a clinical trial and responder analysis. Allergy. 2010 Dec;65(12):1614-21. doi: 10.1111/j.1398-9995.2010.02413.x. PMID 20645937
- [Background] Blumberga G, Groes L, Dahl R. SQ-standardized house dust mite immunotherapy as an immunomodulatory treatment in patients with asthma. Allergy. 2011 Feb;66(2):178-85. doi: 10.1111/j.1398-9995.2010.02451.x. Epub 2010 Sep 30. PMID 20883456
- [Background] Schulze J, Rosewich M, Dressler M, Riemer C, Rose MA, Zielen S. Bronchial allergen challenge using the Medicaid dosimeter. Int Arch Allergy Immunol. 2012;157(1):89-97. doi: 10.1159/000324473. Epub 2011 Sep 7. PMID 21912178
- [Result] Zielen S, Christmann M, Kloska M, Dogan-Yildiz G, Lieb A, Rosewich M, Schubert R, Rose MA, Schulze J. Predicting short term response to anti-inflammatory therapy in young children with asthma. Curr Med Res Opin. 2010 Feb;26(2):483-92. doi: 10.1185/03007990903485148. PMID 20001651
- [Result] Schubert R, Eickmeier O, Garn H, Baer PC, Mueller T, Schulze J, Rose MA, Rosewich M, Renz H, Zielen S. Safety and immunogenicity of a cluster specific immunotherapy in children with bronchial asthma and mite allergy. Int Arch Allergy Immunol. 2009;148(3):251-60. doi: 10.1159/000161585. Epub 2008 Oct 10. PMID 18849616
- [Result] Rosewich M, Schulze J, Eickmeier O, Telles T, Rose MA, Schubert R, Zielen S. Tolerance induction after specific immunotherapy with pollen allergoids adjuvanted by monophosphoryl lipid A in children. Clin Exp Immunol. 2010 Jun;160(3):403-10. doi: 10.1111/j.1365-2249.2010.04106.x. Epub 2010 Mar 16. PMID 20345983